CLINICAL TRIAL: NCT00001570
Title: A Phase I Study of Continuous Intravenous Infusion of PSC 833 and Vinblastine in Patients With Metastatic Renal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970074; 97-C-0074
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Kidney Neoplasms; Neoplasm Metastasis
Keywords: Cytochrome P 450; Multi-Drug Resistance; P-Glycoprotein; Pharmacokinetics
MeSH Terms: conditions — Kidney Neoplasms; Neoplasm Metastasis | interventions — valspodar; Vinblastine

INTERVENTIONS:
Drug: PSC 833
Drug: vinblastine

SUMMARY:
Bolus PSC 833 is administered on Day 1 simultaneously with initiation of 24 hour continuous infusion of PSC 833, followed by another continuous infusion lasting an additional 6 days. To ensure the safety of a 7 day infusion of PSC 833, one patient is treated for 5 days and a second for 6 days, before the first cohort is enrolled.

Vinblastine is administered in escalating doses on days 2-5. At least 3 patients are entered at each dose level. The MTD will be defined as the dose immediately below that at which 2 patients experience dose limiting toxicity.

Treatment continues every 28 days.

DETAILED DESCRIPTION:
The Phase I clinical trial of the combination of 120-hour continuous intravenous infusion of vinblastine with oral PSC 833 has shown activity in patients with advanced malignancies, particularly renal cell cancer. The MTD of vinblastine in combination with the oral drink solution of PSC 833 was determined to be 0.9 mg/m2/day for five days and 12.5 mg/kg po q 12 hours for eight days, respectively. For the soft gel capsule formulation, the MTD was determined to be 0.6 mg/m2/day vinblastine for five days and 4 mg/kg po q 6 hours PSC 833 for eight days. Ataxia was the dose limiting toxicity. Of the 46 patients, two complete remissions and one partial remission were seen among 29 patients with renal cell carcinoma.

In this Phase I study, patients with advanced renal carcinoma will be treated with escalating doses of vinblastine given as a 72 hour infusion, starting at approximately 40% of the total standard dose. A shorter infusion schedule of vinblastine was chosen since there is evidence in other cytotoxic combinations that PSC 833 increases the AUC and decreases the plasma clearance of chemotherapeutic agents by approximately twofold. Cytochrome P 450 3A or CYP3A, which is the major cytochrome enzyme in the metabolism of vinblastine and PSC 833, will be measured during the first and fourth cycle through an in vivo test using a single intravenous dose of midazolam, a short-acting benzodiazepine. Vinblastine and PSC 833 pharmacokinetics will be performed at the same time. For patients with accessible lesions, tumor biopsy will be requested.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically proven renal cancer with clear cell component:

Measurable or evaluable disease;

No brain metastases;

No grade 2 or greater peripheral neuropathy or neurologic toxicity symptoms.

PRIOR/CONCURRENT THERAPY:

Biologic Therapy: Not specified.

Chemotherapy: No prior or concurrent hypersensitivity to PSC 833 or cyclosporine A.

Endocrine Therapy: Not specified.

Radiotherapy: No prior radiation therapy within 4 weeks of study.

Surgery: No major surgery within 4 weeks of study.

Other: No concurrent treatments that interfere with cyclosporine blood concentrations.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance Status: ECOG 0-2.

Life Expectancy: At least 16 weeks.

Hematopoietic:

ANC greater than or equal to 1500/mm(3);

Platelet count greater than or equal to 100,000/mm(3).

Hepatic:

Bilirubin no greater than 1.5 x normal;

AST no greater than 2.5 x normal.

Renal:

Creatinine no greater than 2.0 mg/dL OR;

Creatinine clearance greater than or equal to 50 mL/min.

Cardiovascular:

No concurrent angina or myocardial infarction that has not been appropriately treated.

Other:

Not pregnant or nursing.

Effective contraceptive required of all fertile patients.

Patients with a history of curatively treated basal cell or squamous cell carcinoma are eligible.

No HIV seropositivity.

No chronic hepatitis or cirrhosis.

Patients with concurrent reversible conditions such as diabetes, hypercalcemia, hyperuricemia, hyperviscosity, infection, renal disease, or spinal cord compression are eligible with appropriate therapy.

Patients must give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46
Dates: Start 1997-02; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Chapman AE, Goldstein LJ. Multiple drug resistance: biologic basis and clinical significance in renal-cell carcinoma. Semin Oncol. 1995 Feb;22(1):17-28. No abstract available. PMID 7855615
- [Background] Boote DJ, Dennis IF, Twentyman PR, Osborne RJ, Laburte C, Hensel S, Smyth JF, Brampton MH, Bleehen NM. Phase I study of etoposide with SDZ PSC 833 as a modulator of multidrug resistance in patients with cancer. J Clin Oncol. 1996 Feb;14(2):610-8. doi: 10.1200/JCO.1996.14.2.610. PMID 8636778
- [Background] Twentyman PR. MDR1 (P-glycoprotein) gene expression--implications for resistance modifier trials. J Natl Cancer Inst. 1992 Oct 7;84(19):1458-60. doi: 10.1093/jnci/84.19.1458. No abstract available. PMID 1359150